CLINICAL TRIAL: NCT00387387
Title: An Open-Label, Pharmacokinetic Study of the Safety and Tolerability of Pazopanib in Combination With FOLFOX 6 or CapeOx in Subjects With Colorectal Cancer
Brief Title: Study On Pazopanib When Given With FOLFOX6 (Fluorouracil, Oxaliplatin, Leucovorin) Or CapeOx (Capecitabine, Oxaliplatin)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEG105424
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Neoplasms, Colorectal
Keywords: pharmacokinetics; colorectal cancer; pazopanib; capecitabine; CapeOx; 5-fluorouracil; oxaliplatin; combination therapy; FOLFOX 6
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FOLFOX 6 + Pazopanib (Experimental): Subjects will receive escalating doses of Pazopanib in combination with FOLFOX 6.
  Interventions: Drug: Pazopanib; Drug: FOLFOX 6
- CapeOx + Pazopanib (Experimental): Subjects will receive escalating doses of Pazopanib in combination with CapeOx. CapeOx treatment consisted of IV oxaliplatin (130 mg/m^2) on Day 1 plus oral capecitabine (1000 mg/m^2) twice daily on Days 2 through 14 of every 21-day cycle. Reduced CapeOx treatment was administered according to the same schedule as the CapeOx treatment, but the dose of capecitabine was reduced to 850 mg/m^2 twice daily.
  Interventions: Drug: Pazopanib; Drug: CapeOx

INTERVENTIONS:
Drug: Pazopanib — Pazopanib is an oral inhibitor of vascular endothelial growth factor receptor, platelet-derived growth factor receptor, and c-kit kinases
Drug: FOLFOX 6 — FOLFOX 6 treatment consists of intravenous (IV) oxaliplatin (100 milligram per meter^2[mg/m^2]), and folinic acid (400 mg/m^2), IV 5-fluorouracil bolus (400 mg/m^2) followed by IV 5-fluorouracil (2400 to 3000 mg/m^2) infusion over 48 hours on Day 1 of every 14-day cycle.
  Arms: FOLFOX 6 + Pazopanib
Drug: CapeOx — CapeOx treatment consists of IV oxaliplatin (130 mg/m^2) on Day 1 plus oral capecitabine (1000 mg/m^2) twice daily on Days 2 through 14 of every 21-day cycle. Reduced CapeOx treatment will be administered according to the same schedule as the CapeOx treatment, but the dose of capecitabine will be reduced to 850 mg/m^2 twice daily.
  Arms: CapeOx + Pazopanib

SUMMARY:
This study will test the safety of treating colorectal cancer with a combination of drugs. The current standard treatments of FOLFOX6 or CapeOx will be give in combination with the GSK investigational drug pazopanib.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of locally advanced or metastatic colorectal cancer.
* No prior chemotherapy for metastatic disease.
* Presence of radiologically and/or clinically documented disease.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Adequate bone marrow, hepatic, renal function, Urine Creatinine Ratio (UPC) of <
* A female subject must not be pregnant or breast feeding.
* Able to swallow and retain oral medications.

Exclusion Criteria:

* Has had any major surgery, chemotherapy, hormone therapy, investigational agent, or radiotherapy within the last 28 days
* Prior treatment with pazopanib, or oxaliplatin.
* Known contraindications to the use of oxaliplatin, capecitabine, 5-fluorouracil, or folinic acid.
* Participation in any investigational study within 28 days prior to study treatment.
* Women who are pregnant or lactating.
* Poorly controlled hypertension.
* A history of cardiovascular disease, arrhythmias, or significant ECG abnormalities.
* Any history of stroke.
* Current use of therapeutic warfarin.
* Known brain metastases.
* History of disease significantly affecting gastrointestinal function or major resection of the stomach or small bowel.
* Active infections or other serious illness.
* History of allergy to platinum compounds or heparin.
* Poor venous access.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-10-20 (Actual); Primary Completion 2009-08-14 (Actual); Study Completion 2009-08-14 (Actual)

PRIMARY OUTCOMES:
Plasma AUC(0-24) of pazopanib on Day 1, 14 and 21 Plasma AUC(0-46) of 5-FU and AUC(0-8) of platinum on Day 1 Plasma AUC(0-24) of capecitabine, 5-FU, and platinum on Day 1 | on Day 1, 14 and 21

SECONDARY OUTCOMES:
Pharmacokinetic endpoints (AUC, C24, Cmax, tmax, and half-life)collected predose and 1, 2, 3, 4, 5, 6, 8, and 24 hours on Day 1. Assessment of disease by imaging | collected predose and 1, 2, 3, 4, 5, 6, 8, and 24 hours on Day 1.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- India (2):
  - GSK Investigational Site, Hyderabad, Andhra Pradesh
  - GSK Investigational Site, Pārel
- United Kingdom (3):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Oxford, Oxfordshire
  - GSK Investigational Site, Sutton, Surrey

REFERENCES:
- [Derived] Brady J, Corrie P, Chau I, Digumarti R, Adams LM, Botbyl J, Laubscher KH, Midgley RS, Mallath M. An open-label study of the safety and tolerability of pazopanib in combination with FOLFOX6 or CapeOx in patients with colorectal cancer. Invest New Drugs. 2013 Oct;31(5):1228-35. doi: 10.1007/s10637-013-9938-7. Epub 2013 Feb 28. PMID 23456563
- See also: Results for study VEG105424 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/VEG105424?search=study&study_ids=VEG105424#rs